CLINICAL TRIAL: NCT03827109
Title: Peer Mentoring to Improve Self-management in Youth With IBD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator resignation.
Sponsor: Kelly Boone (Other)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor-Investigator, Kelly Boone, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01NR017533 (NIH)
Record Dates: First submitted 2019-01-14; First posted 2019-02-01 (Actual); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Crohns Disease; Pediatric Ulcerative Colitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Pediatric ulcerative colitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mentoring program (Experimental): The Mentoring Program consists of year-long, 1:1 mentee-mentor relationships with group educational activities, online educational information, and a parent support component. Mentors and mentees are expected to have weekly contact (e.g., text, phone), with in-person contact 1 - 2 times per month. Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. They also provide opportunities to socialize with other mentors and mentees: lunch and games are provided before or after the educational event. Parents participate in a social/support group facilitated by an Investigator while mentees and mentors are socializing. Parents join the mentees and mentors for the educational topics. Due to the COVID-19 pandemic, these activities can be conducted virtually.
  Interventions: Behavioral: Group educational activities; Behavioral: IBD educational website; Behavioral: Monthly check-in calls from program coordinator; Behavioral: Mentor; Behavioral: Fun group activities; Behavioral: Parent support group
- Educational activity program (Active Comparator): The Educational Activity comparison group consists of separate educational group events on the same topics (with no social time), educational information posted online, and monthly encouragement to engage in activities in the community. Due to the COVID-19 pandemic, participants are encouraged to interact socially in safe ways, e.g., outdoors or virtually.
  Interventions: Behavioral: Group educational activities; Behavioral: IBD educational website; Behavioral: Monthly check-in calls from program coordinator

INTERVENTIONS:
Behavioral: Group educational activities — Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. s.
Behavioral: IBD educational website — Website with age-appropriate educational information, including information from the group educational activities.
Behavioral: Monthly check-in calls from program coordinator — Phone calls from coordinator to encourage youth to do something fun with a friend (comparison group) or mentor (Mentoring Program). During the COVID-19 pandemic, virtual activities are encouraged. For those in the Mentoring Program, the coordinator will also ask about the mentee's relationship with the mentor.
Behavioral: Mentor — Mentees will be matched with a mentor for a year-long, 1:1 mentee-mentor relationship. Matching mentors and mentees is based on gender (same), age, geographical proximity, ethnicity, and interests. Mentors and mentees are expected to have weekly contact (e.g., text, phone), with in-person contact 1 - 2 times per month, one of which can be attending a group activity together. Due to the COVID-19 pandemic, a modification was approved so that all study activities can be conducted virtually, e.g., the in-person mentor-mentee monthly activity can be conducted via Skype, and group activities are live streamed
  Arms: Mentoring program
Behavioral: Fun group activities — Program participants vote on "fun" group activities to participate in for support and to learn self-management skills through experiential opportunities and modeling. These are live streamed during the COVID-19 pandemic.
  Arms: Mentoring program
Behavioral: Parent support group — Parents participate in a social/support group facilitated by an Investigator while mentees and mentors are socializing during group events (virtually during the COVID-19 pandemic).
  Arms: Mentoring program

SUMMARY:
This study is a multi-site randomized controlled clinical trial evaluating the efficacy of a peer mentoring program for improving the self-management of youth with IBD. The primary outcomes are youth QOL and functioning in typical life activities. Secondary outcomes are disease outcomes, including disease severity and clinical outcomes (hospital admissions, clinic appointments, missed appointments, procedures). Mentor and parent QOL will also be assessed as secondary outcomes. Mechanisms that may contribute to the effects of the Mentoring Program will be investigated: Parent and child self-efficacy, illness uncertainty, coping, social support and child perceived stigma. Sex will be explored as a moderator.

A total of 200 youth and their parents and 100 mentors will be enrolled. Eligibility criteria for youth include age 10-17 years, parent and child English fluency, and no documented neurodevelopmental disorder or history of hospitalization for a psychiatric or behavioral disorder. Mentors will be ≥16 years, ≥1 year post-diagnosis of IBD and managing their IBD well. They will be rigorously screened via online application, interview, checks of references, driving records, and social media, background check, and successful completion of a 3-hour training. Youth will be randomly assigned to the Mentoring Program or an "Educational Activity" comparison group, with baseline assessments occurring prior to randomization. Follow-up assessments will occur post-intervention and 6 months later.

The Mentoring Program consists of year-long, 1:1 mentee-mentor relationships with group educational activities, online educational information, and a parent support component. Mentors and mentees are expected to have weekly contact (e.g., text, phone), with in-person contact 1 - 2 times per month.

Group activities target self-management skills through experiential opportunities, modeling, and direct instruction. Educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. They also provide opportunities to socialize with other mentors and mentees: lunch and games are provided before or after the educational event.

The Educational Activity comparison group consists of separate educational group events on the same topics (with no social time), educational information posted online, and monthly encouragement to engage in activities in the community.

DETAILED DESCRIPTION:
The proposed study is a multi-site randomized controlled clinical trial evaluating the efficacy of a peer mentoring program for improving the self-management of youth with IBD. The primary outcomes are youth QOL and functioning in typical life activities, which can remain significantly impaired even when the disease is in remission, but have received little empirical attention. Secondary outcomes are disease outcomes, including disease severity and clinical outcomes (hospital admissions, clinic appointments, missed appointments, procedures). Mentor and parent QOL will also be assessed as secondary outcomes. Mechanisms that may contribute to the effects of the Mentoring Program will be investigated: Parent and child self-efficacy, illness uncertainty, coping, social support and child perceived stigma may mediate relationships between mentoring and outcomes. Sex will be explored as a moderator.

A total of 200 youth and their parents and 100 mentors will be enrolled in the study. Eligibility criteria for youth include age 10-17 years, parent and child English fluency, and no documented neurodevelopmental disorder or history of hospitalization for a psychiatric or behavioral disorder. Mentors will be ≥16 years, ≥1 year post-diagnosis of IBD and managing their IBD well. They will be rigorously screened via online application, interview, checks of references, driving records, and social media, background check, and successful completion of a 3-hour training. Youth will be randomly assigned to the Mentoring Program or an "Educational Activity" comparison group, with baseline assessments occurring prior to randomization. Follow-up assessments will occur post-intervention and 6 months later. Youth in the Educational Activity group will be yoked to those in Mentoring Program, and the timing of their follow-up assessments will correspond to their yoked peer.

The Mentoring Program was developed via focus groups, an NIH-funded pilot study, national mentoring resources, and the PI's 10 years of experience with Big Brothers Big Sisters. It consists of year-long, 1:1 mentee-mentor relationships with group educational activities, online educational information, and a parent support component. Matching mentors and mentees is based on gender (same), age, geographical proximity, ethnicity, and interests. Mentors and mentees are expected to have weekly contact (e.g., text, phone), as well as participate in an activity (in person or virtually) 1 - 2 times per month, one of which can be attending a group activity together. The investigators expect the relationship to last 1 year, which is associated with better outcomes than shorter relationships.

Group activities target self-management skills through experiential opportunities, modeling, and direct instruction. Educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area (e.g., dietitian, pediatric gastroenterologists). They also provide opportunities to socialize with other mentors and mentees: lunch and games are provided before or after the educational event. Parents in the Mentoring Program participate in a social/support group facilitated by an Investigator while mentees and mentors are socializing. Parents join the mentees and mentors for the educational topics.

The Educational Activity comparison group consists of separate educational group events on the same topics (with no social or support time), educational information posted online, and monthly encouragement to engage in activities in the community.

Due to the COVID-19 pandemic, a modification was approved so that all study activities can be conducted virtually, e.g., the in-person mentor-mentee monthly activity can be conducted via Skype, and group activities are live streamed.

ELIGIBILITY:
Inclusion Criteria:

Mentees:

* Diagnosis of IBD
* Age 10 - 17 years
* Parent and child English fluency
* No documented neuro-developmental disorder or history of hospitalization for a psychiatric or behavioral disorder

Mentors:

* ≥16 years
* ≥1 year post-diagnosis of IBD
* Managing their IBD well
* Pass a screening that includes an online application, interview, 3 character references, checks of driving records and social media, background check, mentor training

Exclusion Criteria:

Mentees: No documented neuro-developmental disorder or history of hospitalization for a psychiatric or behavioral disorder

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Abigail Wexner Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be archived with the digital repository of the Inter-university Consortium for Political and Social Research (ICPSR). NCH is a member of ICPSR via the Ohio State University; thus ICPSR can curate the data using funds provided by membership dues. ICPSR can archive the full dataset and its documentation, supporting the data through future changing technologies, new media, and data formats. ICPSR will make the data available to the broader research community via files that may be accessed directly via the ICPSR Web site. Approximately 776 universities, government agencies, and other institutions are members of ICPSR. Member institutions have full direct access to ICPSR's data archives and to all of ICPSR's services and can download the data. Non-members may purchase the files. The data will be deposited with the repository at the completion of the study and disseminated in one year to give the investigators time to publish their findings.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be deposited with the repository at the completion of the study but not disseminated for one year to give the investigators time to publish their findings.
Access Criteria: Users with an ICPSR MyData account and an authorized IP address from a member institution may download the data, and non-members may purchase the files.

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After recruitment, parents and youth will complete measures at baseline. Data will be collected in participants' homes to reduce the number of hospital visits required for families. Then they will be randomized into the mentoring program or comparison group.
Groups:
- Mentoring Program (Child): The Mentoring Program consists of year-long, 1:1 mentee-mentor relationships with group educational activities, online educational information, and a parent support component. Mentors and mentees are expected to have weekly contact (e.g., text, phone), with in-person contact 1 - 2 times per month. Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. They also provide opportunities to socialize with other mentors and mentees: lunch and games are provided before or after the educational event. Parents participate in a social/support group facilitated by an Investigator while mentees and mentors are socializing. Parents join the mentees and mentors for the educational topics.
- Educational Activity Program (Child): The Educational Activity comparison group consists of separate educational group events on the same topics (with no social time), educational information posted online, and monthly encouragement to engage in activities in the community. Due to the COVID-19 pandemic, participants are encouraged to interact socially in safe ways, e.g., outdoors or virtually.
  Group educational activities: Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. s.
  IBD educational website: Website with age-appropriate educational information, including information from the group educational activities.
  Monthly check-in calls from program coordinator: Phone calls from coordinator to encourage youth to do something fun with a friend (comparison group) or mentor (Mentoring Program). During the COVID-19 pandemic, virtual activities are encouraged. For those in the Mentoring Program, the coordinator will also ask about the mentee's relationship with the mentor.
- Mentoring Program (Parent): The Mentoring Program consists of year-long, 1:1 mentee-mentor relationships with group educational activities, online educational information, and a parent support component. Mentors and mentees are expected to have weekly contact (e.g., text, phone), with in-person contact 1 - 2 times per month. Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. They also provide opportunities to socialize with other mentors and mentees: lunch and games are provided before or after the educational event. Parents participate in a social/support group facilitated by an Investigator while mentees and mentors are socializing. Parents join the mentees and mentors for the educational topics. Due to the COVID-19 pandemic, these activities can be conducted virtually.
- Educational Activity Program (Parent): The Educational Activity comparison group consists of separate educational group events on the same topics (with no social time), educational information posted online, and monthly encouragement to engage in activities in the community. Due to the COVID-19 pandemic, participants are encouraged to interact socially in safe ways, e.g., outdoors or virtually.
  Group educational activities: Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area.
  IBD educational website: Website with age-appropriate educational information, including information from the group educational activities.
  Monthly check-in calls from program coordinator: Phone calls from coordinator to encourage youth to do something fun with a friend (comparison group) or mentor (Mentoring Program). During the COVID-19 pandemic, virtual activities are encouraged. For those in the Mentoring Program, the coordinator will also ask about the mentee's relationship with the mentor.
- Mentors: Mentors will facilitate group educational and socialization activities for children assigned to the mentorship program arm. Parents assigned to the mentorship program arm will join the mentors and mentees for educational topics.
Period: Overall Study
Arm/Group | Mentoring Program (Child) | Educational Activity Program (Child) | Mentoring Program (Parent) | Educational Activity Program (Parent) | Mentors
Started | 55 | 56 | 55 | 56 | 63
Completed | 40 | 39 | 0 | 0 | 0
Not Completed | 15 | 17 | 55 | 56 | 63

BASELINE CHARACTERISTICS:
Groups:
- Mentoring Program (Child); Mentoring Program (Parent): The Mentoring Program consists of year-long, 1:1 mentee-mentor relationships with group educational activities, online educational information, and a parent support component. Mentors and mentees are expected to have weekly contact (e.g., text, phone), with in-person contact 1 - 2 times per month. Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area. They also provide opportunities to socialize with other mentors and mentees: lunch and games are provided before or after the educational event. Parents participate in a social/support group facilitated by an Investigator while mentees and mentors are socializing. Parents join the mentees and mentors for the educational topics. Due to the COVID-19 pandemic, these activities can be conducted virtually.
- Educational Activity Program (Child); Educational Activity Program (Parent): The Educational Activity comparison group consists of separate educational group events on the same topics (with no social time), educational information posted online, and monthly encouragement to engage in activities in the community. Due to the COVID-19 pandemic, participants are encouraged to interact socially in safe ways, e.g., outdoors or virtually.
  Group educational activities: Group educational topics include nutrition, stress, IBD and school, and disease management, and are taught by experts in each content area.
  IBD educational website: Website with age-appropriate educational information, including information from the group educational activities.
  Monthly check-in calls from program coordinator: Phone calls from coordinator to encourage youth to do something fun with a friend (comparison group) or mentor (Mentoring Program). During the COVID-19 pandemic, virtual activities are encouraged. For those in the Mentoring Program, the coordinator will also ask about the mentee's relationship with the mentor.
- Total: Total of all reporting groups
Arm/Group | Mentoring Program (Child) | Educational Activity Program (Child) | Mentoring Program (Parent) | Educational Activity Program (Parent) | Mentors | Total
Number analyzed (Participants) | 55 | 56 | 55 | 56 | 63 | 285
Age, Customized [Mean (Standard Deviation); unit: Years] — Population: 3 Mentors' age data missing; Only participant age data from Children and Mentors was collected in this study.
  Years
    Participant Age: number analyzed (Participants) | 55 | 56 | 0 | 0 | 60 | 171
    Participant Age | 11.8 (1.6) | 12.2 (2.0) |  |  | 21 (5.1) | 12.7 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 55 | 56 | 46 | 204
  Male | 30 | 34 | 0 | 0 | 17 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data related to participant race within each arm was not recorded until later time point.
  Participants
    American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
    Asian | 2 | 1 | 2 | 1 | 3 | 9
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 7 | 6 | 7 | 6 | 4 | 30
    White | 38 | 47 | 39 | 43 | 54 | 221
    More than one race | 7 | 2 | 1 | 1 | 2 | 13
    Unknown or Not Reported | 0 | 0 | 6 | 5 | 0 | 11
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 55 | 56 | 63 | 285

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Youth Quality of Life: PedsQL
Description: PedsQL (full, unabbreviated scale name). Construct: Youth quality of life. Scores range from 0-100 with higher scores indicating higher quality of life. Total score will be used.
Time Frame: 12 months post mentor-mentee introduction
Population: 0 participants analyzed due to early study termination. Study was terminated before data was collected, so no data was collected to analyze. Due to complications from the COVID-19 epidemic, research procedures related to data collection and analysis were significantly impacted and thus data collection/analysis did not occur before study closure.
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

2. Primary Outcome: 18 Month Youth Quality of Life: PedsQL
Description: as for outcome 1
Time Frame: 18 months post mentor-mentee introduction
Population: 0 participants analyzed due to early study termination. Study was terminated before data was collected, so no data was collected to analyze. Due to complications from the COVID-19 epidemic, research procedures related to data collection/analysis were significantly impacted and thus data collection/analysis did not occur before study closure.
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

3. Primary Outcome: 12 Month Change From Baseline Youth Quality of Life: PedsQL
Description: as for outcome 1
Time Frame: Baseline to 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

4. Primary Outcome: 18 Month Change From Baseline Youth Quality of Life: PedsQL: Physical
Description: Pediatric Quality of Life Inventory (PedsQL), Physical Domain (full, unabbreviated scale name). Construct: Youth quality of life. Scores range from 0-100 with higher scores indicating higher quality of life. Total score will be used. Score below reflects change from baseline to 18-months post mentor-mentee introduction, with higher absolute values reflecting greater change.
Time Frame: Baseline to 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

5. Primary Outcome: 12 Month Youth Functional Disability
Description: Functional Disability Inventory. Assess adaptive functioning in every day life. Scores range from 0 - 60 with higher scores indicating greater disability. Total score will be used.
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

6. Primary Outcome: 18 Month Youth Functional Disability
Description: as for outcome 5
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

7. Primary Outcome: 12 Month Change From Baseline Youth Functional Disability
Description: as for outcome 5
Time Frame: Baseline to 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

8. Primary Outcome: 18 Month Change From Baseline Youth Functional Disability
Description: as for outcome 5
Time Frame: Baseline to 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

9. Secondary Outcome: 12 Month Youth Disease Outcomes - Crohn's Disease Severity
Description: Disease severity: Pediatric Crohn's Disease Activity Index total score. A standard measure of disease severity that is comprised of information obtained from patient recall (pain severity, stool frequency, limitation of activities), examination (weight, height, abdominal tenderness, perirectal disease, extra- intestinal manifestations), and laboratory data. The Pediatric Crohn's Disease Activity Index total score will be used. Higher scores indicate more severe disease.
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

10. Secondary Outcome: 12 Month Youth Disease Outcomes - Ulcerative Colitis Severity
Description: Disease severity: Pediatric Ulcerative Colitis Activity Index total score. A standard Pediatric Ulcerative Colitis Activity Index. a standard measure of disease severity that is comprised pain severity, stool frequency and consistency, rectal bleeding, nocturnal bowel movements, and limitation of activities. The Pediatric Ulcerative Colitis Activity Index total score will be used. Higher scores indicate more severe disease.
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

11. Secondary Outcome: 18 Month Youth Disease Outcomes - Crohn's Disease Severity
Description: as for outcome 9
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

12. Secondary Outcome: 18 Month Youth Disease Outcomes - Ulcerative Colitis Severity
Description: as for outcome 10
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

13. Secondary Outcome: 12 Month Number of Hospital Admissions in Previous 6 Months
Description: 12 month number of hospital admissions in previous 6 months
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

14. Secondary Outcome: 18 Month Number of Hospital Admissions in Previous 6 Months
Description: 18 month number of hospital admissions in previous 6 months
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

15. Secondary Outcome: 12 Month Number of Clinic Appointments in Previous 6 Months
Description: 12 month number of clinic appointments in previous 6 months
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

16. Secondary Outcome: 18 Month Number of Clinic Appointments in Previous 6 Months
Description: 18 month number of clinic appointments in previous 6 months
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

17. Secondary Outcome: 12 Month Number of Missed Appointments in Previous 6 Months
Description: 12 month number of missed appointments in previous 6 months
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

18. Secondary Outcome: 18 Month Number of Missed Appointments in Previous 6 Months
Description: 18 month number of missed appointments in previous 6 months
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

19. Secondary Outcome: 12 Month Number of Procedures in Previous 6 Months
Description: 12 month number of procedures appointments in previous 6 months
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

20. Secondary Outcome: 18 Month Number of Procedures in Previous 6 Months
Description: 18 month number of procedures appointments in previous 6 months
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

21. Secondary Outcome: 12 Months Mentor QOL
Description: PedsQL Adult Report (full, unabbreviated scale name). Construct: Mentor quality of life. Scores range from 0-100 with higher scores indicating higher quality of life. Total score will be used.
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentoring Program | Educational Activity Program
Number analyzed (Participants) | 0 | 0
Participants | 0 | 0

22. Secondary Outcome: 18 Months Mentor QOL
Description: as for outcome 21
Time Frame: 18 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Mentors: Mentors paired with participants in the mentoring treatment group.
Arm/Group | Mentors
Number analyzed (Participants) | 0
Participants | 0

23. Secondary Outcome: 12 Month Change From Baseline Mentor QOL
Description: as for outcome 21
Time Frame: Baseline to 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Mentors
Number analyzed (Participants) | 0
Participants | 0

24. Secondary Outcome: 12 Month Parent QOL
Description: PedsQL Family Impact Module (full, unabbreviated scale name). Construct: Parent quality of life and the impact a child's chronic illness has on the family. Scores range from 0-100 with higher scores indicating higher quality of life. Total score will be used.
Time Frame: 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Parents: Parents of children enrolled in the Mentoring or Comparison treatment arm.
Arm/Group | Parents
Number analyzed (Participants) | 0
Participants | 0

25. Secondary Outcome: 12 Month Change From Baseline Parent QOL
Description: as for outcome 24
Time Frame: Baseline to 12 months post mentor-mentee introduction
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Parents
Number analyzed (Participants) | 0
Participants | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Mentoring Program (Child) | Educational Activity Program (Child) | Mentoring Program (Parent) | Educational Activity Program (Parent) | Mentors
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56 | 0/55 | 0/56 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 0/55 | 0/56 | 0/63
Other Adverse Events (participants affected / at risk) | 7/55 | 5/56 | 0/55 | 0/56 | 0/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mentoring Program (Child) (N=55) | Educational Activity Program (Child) (N=56) | Mentoring Program (Parent) (N=55) | Educational Activity Program (Parent) (N=56) | Mentors (N=63)
COVID-19 (Infections and infestations) | 5 (8) | 3 (3) | NA | NA | NA
Worsening IBD Symptoms (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA | NA | NA
Other Illness (Infections and infestations) | 3 (3) | 2 (2) | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT03827109/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT03827109/ICF_001.pdf